CLINICAL TRIAL: NCT06180837
Title: Biomarkers of Habitual Short Sleep and Related Cardiometabolic Risk
Brief Title: Effect of Sleep Extension on Ceramides in People with Overweight and Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Depner, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 164764
Record Dates: First submitted 2023-11-14; First posted 2023-12-26 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Lifestyle Factors; Overweight and Obesity; Insulin Sensitivity; Eating Habit; Sleep Hygiene; Type 2 Diabetes; Sleep; Sleep Deprivation; Insufficient Sleep Syndrome
Keywords: sleep; insulin sensitivity
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Feeding Behavior; Sleep Hygiene; Diabetes Mellitus, Type 2; Sleep Deprivation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Group allocation will be blinded to research staff and participants until the conclusion of the baseline segment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Provided with general health information on diet and physical activity.
- Intervention Group (Experimental): Sleep extension-based intervention focused on increasing time in bed by 2 hours per night.
  Interventions: Behavioral: Sleep Extension Intervention

INTERVENTIONS:
Behavioral: Sleep Extension Intervention — Sleep extension-based intervention focused on increasing time spent in bed by 2 hours per night by directly scheduling assigned bed and waketimes based on participant's individual schedules. Participants will receive weekly sleep tips and counseling on improving their sleep duration.
  Arms: Intervention Group

SUMMARY:
The overall goal is to determine how a sleep extension intervention (increasing time in bed) in individuals who maintain less than 6.5 hours sleep per night affects their plasma ceramides and insulin sensitivity. Participants will undergo a randomized controlled trial, with sleep extension (intervention) and healthy lifestyle (control) groups. The sleep extension is designed to increase participant's time in bed by 2 hours per night. Alternatively, the control group will receive basic health information (e.g., physical activity, goal setting, and nutrition when eating out).

DETAILED DESCRIPTION:
A randomized controlled trial with real-world sleep extension in adults with overweight and obesity who habitually obtain short sleep duration will be conducted. Group allocation will be 1:1 and research staff and participants will be blinded until the conclusion of the baseline segment. The sleep extension group will receive counseling and instruction to increase nightly time in bed by 2 hours per night. Participants randomized to control will maintain their habitual sleep habits in their home environment. The intervention segment will last 8 weeks regardless of group assignment. Both groups will have equal contact time with the study team.

Prior to enrollment participants will complete a clinical overnight sleep disorders screening. Baseline consists of an ~1-week ambulatory real-world monitoring segment. Following baseline, participants will be randomized 1:1 to either the sleep extension or control group for 8 weeks at home (intervention segment). Throughout the study, sleep duration will be monitored using an actiwatch wrist-device and a daily electronic sleep log. Following the baseline and intervention segments participants will complete rigorous overnight laboratory visits to assess plasma ceramides (targeted metabolomics assay) and insulin sensitivity (hyperinsulinemic-euglycemic clamp).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-45 years old; equal numbers of men and women
2. Body mass index (BMI): 27.5-34.9 kg/m2
3. Sleep Habits: habitual self-reported average total sleep time (TST) <6.5 hours per night for prior 6 months

Exclusion Criteria:

1. Clinically diagnosed sleep disorder or major psychiatric illness
2. Evidence of significant organ dysfunction or disease (e.g., heart disease, kidney disease)
3. Clinically diagnosed diabetes or fasting plasma glucose ≥126 mg/dL or HbA1c ≥6.5%
4. Use of prescription drugs or substances known to influence sleep or glucose metabolism, or anticoagulant medications.
5. Cancer that has been in remission less than 5 years
6. Pregnant/nursing, experiencing menopause or post-menopausal
7. Shift-work: current or history of within last year
8. Weight change: >10% of body weight over prior six months
9. Current enrollment in weight loss or physical activity program like the Diabetes Prevention Program
10. Currently smoking
11. Alcohol intake>14 drinks per week or >3 drinks per day

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Total Plasma Ceramides | Immediately after the intervention
  Total plasma ceramides will be measured by assessing plasma ceramides by targeted metabolomics.
Insulin Sensitivity | Immediately after the intervention
  Insulin sensitivity will be measured by the glucose infusion rate per kg body weight during the hyperinsulinemic-euglycemic clamp.

SECONDARY OUTCOMES:
Average (per week) nightly total sleep time (change from baseline) | Analyzed as change from baseline for each week of the ~8 week experimental segment
  Wrist-actigraphy
Average (per week) sleep satisfaction change from baseline | Analyzed as change from baseline for each week of the ~8 week experimental segment
  5 point likert scale on daily sleep log (1 = very good; 5 = very poor)
Average (per week) timing of food intake change from baseline | During the baseline ambulatory assessment and weeks 2, 4, 6, and 8 of the intervention ambulatory assessment.
  Time of day 50% of calories are consumed collected by picture based food diaries. Average per week will consist of two weekdays and one weekend day
Average (per week) daytime alertness change from baseline | Time Frame: Analyzed as change from baseline for each week of the ~8 week experimental segment
  5 point likert scale on daily sleep log (1= most alert; 5 = not alert at all)
Individual C16, C18, C20, C22, C24, and C24:1 Plasma Ceramides, Dihydroceramides, Glucosylceramides, and fourteen Sphingolipids. | Immediately after the intervention
  Targeted metabolomics assay, 32 total metabolites.
Circadian Phase (change from baseline) | Immediately after the intervention
  dim-light melatonin onset quantified from salivary melatonin samples
Body Mass Index | Immediately after the intervention
  Nurses will collect height and body weight using standard procedures.
Cardiac Event Risk Test 1 (CERT 1) | Immediately after the intervention
  The Cardiac Event Risk Test 1 (CERT1) is used to evaluate the risk of major adverse cardiovascular events and can be calculated using data from our targeted metabolomics assay. The scale is from 0-12, 0 being the lowest risk and 12 being the highest level of risk.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Health Research Complex--University of Utah, Salt Lake City, Utah, United States